

## Croydon University Hospital 530 London Road

530 London Road Croydon CR7 7YE

Switchboard Tel: (020) 8401 3000

## Women & Children's Directorate

Direct Line Tel: (020) 8401 3161 Direct Fax: (020) 8401 3681

Email: abdul.sultan@croydonhealth.nhs.uk

**Informed Consent Form** 

| Study Nui | mber: | | | |
|---|---|---|---|---|
| ECHO – Effect of Copper on the Healing of Obstetric wounds | | | | |
| | | | Please sig | n the box with initials |
| sh | onfirm that I have read<br>eet, dated 21/09/2015<br>e opportunity to ask qu | , for the above st | | |
| fre | I understand that my participation is voluntary and that I am free to withdraw at any time without giving any reason and without my medical care or legal rights being affected. | | | |
| at<br>my | 3. I understand that sections of my medical notes may be looked at by responsible individuals in this study where it is relevant to my taking part in research. I give permission to these individuals to have access to my records. | | | |
| | I consent for my GP to be informed about my participation in this study. | | | |
| 5. la | gree to take part in th | is study. | | |
| Name of p | patient | Date | Signature | |
| Name of researcher Date Sign | | Signature | | |